CLINICAL TRIAL: NCT05541120
Title: Effect of Remote Patient Monitoring and Patient Education on Patient Activation and Glycemic Control in Individuals With Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants eligible for study
Sponsor: Tracy Jalbuena MD (Other)
Collaborators: MaineHealth (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Tracy Jalbuena MD, Clinical Lead for Telehealth, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00000
Record Dates: First submitted 2022-08-30; First posted 2022-09-15 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: remote patient monitoring; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial of the use of RPM compared to usual care among MaineHealth's rural patients with poorly controlled diabetes, where the participant's diabetes is managed primarily by primary care (as opposed to endocrinology). Usual care is defined as participation in Living Well with Diabetes/Virtual Diabetes Self-Management Program, PCP evaluation and management at the providers' discretion, including medication adjustment or interventions, and other types of interventions depending on clinical judgement. This may include eConsults between the provider and a pharmacist, in-person visits between the provider and the patient, synchronous telemedicine visits between the provider and the patient, and synchronous telemedicine visits between the pharmacist and the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living Well with Diabetes (No Intervention): Usual care is defined as participation in Living Well with Diabetes/Virtual Diabetes Self-Management Program, PCP evaluation and management, including medication adjustment or interventions, and other types of interventions depending on clinical judgement. This may include eConsults between the provider and a pharmacist, in-person visits between the provider and the patient, synchronous telemedicine visits between the provider and the patient, and synchronous telemedicine visits between the pharmacist and the patient.
- Living Well with Diabetes + Remote Patient Monitoring (Experimental): Remote patient monitoring as the intervention is defined as a tablet and Bluetooth-enabled glucometer technology that collects point-of-care (POC) blood glucose data from a patient outside of a traditional clinical setting, and securely transmits this data to Epic for review and potential intervention.
  Interventions: Device: Remote Patient Monitoring

INTERVENTIONS:
Device: Remote Patient Monitoring — Remote patient monitoring as the intervention is defined as a tablet and Bluetooth-enabled glucometer technology that collects point-of-care (POC) blood glucose data from a patient outside of a traditional clinical setting, and securely transmits this data to Epic for review and potential intervention.
  Arms: Living Well with Diabetes + Remote Patient Monitoring

SUMMARY:
This is a randomized controlled trial of the use of Remote Patient Monitoring (RPM) compared to usual care among rural patients with poorly controlled type 2 diabetes. Usual care is defined as participation in Living Well with Diabetes/Virtual Diabetes Self-Management Program and Primary Care Provider evaluation and management at the providers' discretion, including medication adjustment or interventions, and other types of interventions depending on clinical judgement.

DETAILED DESCRIPTION:
Effect of Remote Patient Monitoring and Patient Education on Patient Activation and Glycemic Control in Individuals with Type 2 Diabetes

Summary

ABSTRACT

In 2021, the MaineHealth Telehealth team was awarded a five-year, $1.7 million "Evidence-Based Telehealth Network Program" grant (EB TNPG) from Health Resources and Services Administration (HRSA). This grant is aimed at improving patient access to educational and management services for patients with type 2 diabetes in the rural Maine primary care setting by implementing RPM. The RPM devices will be used to transmit a participant's home point-of-care blood glucose values directly into MaineHealth's electronic medical record in real time. While there is strong evidence for diabetes self-management programs such as Living Well with Diabetes, the importance of patient engagement in clinical outcomes, the validity of the Patient Activation Measure (PAM-13®) survey to measure patient activation, and the overall efficacy of remote patient monitoring, there have been no randomized controlled trials looking at patient activation in remote patient monitoring in this important patient group. The investigators aim to address this in this study by conducting a randomized controlled trial of the use of RPM among rural patients with poorly controlled type 2 diabetes. The control group will have usual primary care provider care, including patient self-management tools, while the intervention group will have usual care + RPM.

The investigators hypothesize that participation in RPM will be associated with decreases in HbA1c, increases in patient activation as measured by PAM-13® survey, and that increases in patient activation will be associated with decreases in HbA1c.

STUDY PROCESS

The study will be conducted over 5 years, and participants will be enrolled on a continuous rolling basis, with 70 total RPM kits available at any one time from a 3rd party vendor, Health Recovery Solutions (HRS). The maximum total number of participants the study can accommodate is 700, with 350 participants in each arm. The study team hopes for total enrollment as close to 700 as possible, but understands that total enrollment may be significantly less than 700. Point-of-care blood glucose values from the RPM study arm will flow into MaineHealth's electronic medical record (Epic) in real time. Every other week, the values will be reviewed by a clinical pharmacist with expertise in diabetes management. If an intervention or adjustment in the patient's regimen is indicated, the pharmacist will reach out to the Primary Care Provider (PCP) team to make this recommendation. The RPM intervention for each participant will be 6 months, at which point HRS will collect the RPM electronic tablet, and the PAM-13® survey will be administered. At 9 months after enrollment, the third HbA1c value will be collected from the electronic medical record, and the third administration of PAM-13® will take place.

The PAM-13® survey will be administered through one of two methods 1) REDCap electronic form, the link for which will be sent to the participant by email, or 2) by telephone, administered by the Study Coordinator.

Recruitment of participants will continue through the early part of 2026. Data will be analyzed during spring and summer of 2026, and the grant's end date is August 31, 2026.

This study has been approved by MaineHealth's IRB as of Aug 5, 2022.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in Living Well with Diabetes education program
* Have an HbA1c% ≥ 8 in the prior 6 months
* Be capable of providing consent
* Be adults (age 18 or over)

Exclusion Criteria:

* Primarily managed by endocrinology for their diabetes (> 1 visit with endocrinology in the previous 12 months)
* Incarcerated
* PCP not at one of the 30 primary care practices listed (see attachment List of PCP Practices)
* Diagnosed with type 1 diabetes
* Candidate for continuous glucose monitoring, as defined by Centers for Medicare and Medicaid Services as using at least three insulin injections per day, any combination of types of insulins
* Pregnant
* Have previously participated in the Living Well with Diabetes/Virtual Diabetes Self-Management Program
* Have previously used a remote patient monitoring device for diabetes management
* Have a diagnosis of dementia or other clinical diagnosis that would impair participation capacity
* Currently participating in any other clinical trial regarding diabetes care or management
* Currently enrolled in hospice
* Currently residing in a long term care or rehabilitation facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean HbA1c% | 6 months after enrollment
  Average glycated hemoglobin
Mean HbA1c% | 9 months after enrollment
  Average glycated hemoglobin
Mean change in HbA1c% | 6 months after enrollment
  Average change in percentage of HbA1c from baseline to 6 months after enrollment
Mean change in HbA1c% | 9 months after enrollment
  Average change in percentage of HbA1c from baseline to 9 months after enrollment
Percentage of participants in each group who have HbA1c < 7% | 6 months after enrollment
  Percentage of participants in each group with HbA1c < 7%
Percentage of participants in each group who have HbA1c < 7% | 9 months after enrollment
  Percentage of participants in each group with HbA1c < 7%

SECONDARY OUTCOMES:
PAM-13 at 6 months after enrollment | 6 months after enrollment
  PAM-13 Patient Activation Measure Survey
  Unabbreviated scale title: Patient Activation Measure 13-Item Survey Minimum value: 0 Maximum value: 100 Higher values are associated with better health outcomes
PAM-13 at 9 months after enrollment | 9 months after enrollment
  PAM-13 Patient Activation Measure Survey
  PAM-13 Patient Activation Measure Survey
  Unabbreviated scale title: Patient Activation Measure 13-Item Survey Minimum value: 0 Maximum value: 100 Higher values are associated with better health outcomes
Mean change in PAM-13 at 6 months | 6 months after enrollment
  Average change in PAM-13 Patient Activation Measure Survey score from baseline to 6 months after enrollment
  Unabbreviated scale title: Patient Activation Measure 13-Item Survey Minimum value: 0 Maximum value: 100 Higher values are associated with better health outcomes
Mean change in PAM-13 at 9 months | 9 months after enrollment
  Average change in PAM-13 Patient Activation Measure Survey score from baseline to 9 months after enrollment
  Unabbreviated scale title: Patient Activation Measure 13-Item Survey Minimum value: 0 Maximum value: 100 Higher values are associated with better health outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Jalbuena, MD, Principal Investigator — MaineHealth
Locations (1):
- PenBay Medical Center, Rockport, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almutairi N, Hosseinzadeh H, Gopaldasani V. The effectiveness of patient activation intervention on type 2 diabetes mellitus glycemic control and self-management behaviors: A systematic review of RCTs. Prim Care Diabetes. 2020 Feb;14(1):12-20. doi: 10.1016/j.pcd.2019.08.009. Epub 2019 Sep 20. PMID 31543458
- [Background] American Diabetes Association. Economic Costs of Diabetes in the U.S. in 2017. Diabetes Care. 2018 May;41(5):917-928. doi: 10.2337/dci18-0007. Epub 2018 Mar 22. PMID 29567642
- [Background] Andersen JA, Scoggins D, Michaud T, Wan N, Wen M, Su D. Racial Disparities in Diabetes Management Outcomes: Evidence from a Remote Patient Monitoring Program for Type 2 Diabetic Patients. Telemed J E Health. 2021 Jan;27(1):55-61. doi: 10.1089/tmj.2019.0280. Epub 2020 Apr 17. PMID 32302521
- [Background] Bahrom NH, Ramli AS, Isa MR, Baharudin N, Badlishah-Sham SF, Mohamed-Yassin MS, Abdul-Hamid H. Validity and reliability of the Patient Activation Measure(R) (PAM(R))-13 Malay version among patients with Metabolic Syndrome in primary care. Malays Fam Physician. 2020 Nov 10;15(3):22-34. eCollection 2020. PMID 33329860
- [Background] Bomba F, Markwart H, Muhlan H, Menrath I, Ernst G, Thyen U, Schmidt S. Adaptation and validation of the German Patient Activation Measure for adolescents with chronic conditions in transitional care: PAM(R) 13 for Adolescents. Res Nurs Health. 2018 Feb;41(1):78-87. doi: 10.1002/nur.21831. Epub 2017 Dec 20. PMID 29266283
- [Background] Boren SA, Fitzner KA, Panhalkar PS, Specker JE. Costs and benefits associated with diabetes education: a review of the literature. Diabetes Educ. 2009 Jan-Feb;35(1):72-96. doi: 10.1177/0145721708326774. PMID 19244564
- [Background] Boyle JP, Thompson TJ, Gregg EW, Barker LE, Williamson DF. Projection of the year 2050 burden of diabetes in the US adult population: dynamic modeling of incidence, mortality, and prediabetes prevalence. Popul Health Metr. 2010 Oct 22;8:29. doi: 10.1186/1478-7954-8-29. PMID 20969750
- [Background] Brenk-Franz K, Hibbard JH, Herrmann WJ, Freund T, Szecsenyi J, Djalali S, Steurer-Stey C, Sonnichsen A, Tiesler F, Storch M, Schneider N, Gensichen J. Validation of the German version of the patient activation measure 13 (PAM13-D) in an international multicentre study of primary care patients. PLoS One. 2013 Sep 30;8(9):e74786. doi: 10.1371/journal.pone.0074786. eCollection 2013. PMID 24098669
- [Background] Chrvala CA, Sherr D, Lipman RD. Diabetes self-management education for adults with type 2 diabetes mellitus: A systematic review of the effect on glycemic control. Patient Educ Couns. 2016 Jun;99(6):926-43. doi: 10.1016/j.pec.2015.11.003. Epub 2015 Nov 22. PMID 26658704
- [Background] Cunha CM, da Cunha DCPT, Manzato RO, Nepomuceno E, da Silva D, Dantas RAS. Validation of the Brazilian Version of the Patient Activation Measure 13. J Nurs Meas. 2019 Apr 1;27(1):97-113. doi: 10.1891/1061-3749.27.1.97. PMID 31068494
- [Background] Dieleman JL, Baral R, Birger M, Bui AL, Bulchis A, Chapin A, Hamavid H, Horst C, Johnson EK, Joseph J, Lavado R, Lomsadze L, Reynolds A, Squires E, Campbell M, DeCenso B, Dicker D, Flaxman AD, Gabert R, Highfill T, Naghavi M, Nightingale N, Templin T, Tobias MI, Vos T, Murray CJ. US Spending on Personal Health Care and Public Health, 1996-2013. JAMA. 2016 Dec 27;316(24):2627-2646. doi: 10.1001/jama.2016.16885. PMID 28027366
- [Background] Egede LE, Williams JS, Voronca DC, Knapp RG, Fernandes JK. Randomized Controlled Trial of Technology-Assisted Case Management in Low Income Adults with Type 2 Diabetes. Diabetes Technol Ther. 2017 Aug;19(8):476-482. doi: 10.1089/dia.2017.0006. Epub 2017 Jun 5. PMID 28581821
- [Background] Fowles JB, Terry P, Xi M, Hibbard J, Bloom CT, Harvey L. Measuring self-management of patients' and employees' health: further validation of the Patient Activation Measure (PAM) based on its relation to employee characteristics. Patient Educ Couns. 2009 Oct;77(1):116-22. doi: 10.1016/j.pec.2009.02.018. Epub 2009 Apr 7. PMID 19356881
- [Background] Glasgow RE, Wagner EH, Schaefer J, Mahoney LD, Reid RJ, Greene SM. Development and validation of the Patient Assessment of Chronic Illness Care (PACIC). Med Care. 2005 May;43(5):436-44. doi: 10.1097/01.mlr.0000160375.47920.8c. PMID 15838407
- [Background] Greene J, Hibbard JH. Why does patient activation matter? An examination of the relationships between patient activation and health-related outcomes. J Gen Intern Med. 2012 May;27(5):520-6. doi: 10.1007/s11606-011-1931-2. PMID 22127797
- [Background] Haas L, Maryniuk M, Beck J, Cox CE, Duker P, Edwards L, Fisher EB, Hanson L, Kent D, Kolb L, McLaughlin S, Orzeck E, Piette JD, Rhinehart AS, Rothman R, Sklaroff S, Tomky D, Youssef G; 2012 Standards Revision Task Force. National standards for diabetes self-management education and support. Diabetes Care. 2014 Jan;37 Suppl 1(Suppl 1):S144-53. doi: 10.2337/dc14-S144. No abstract available. PMID 24357210
- [Background] Hellstrom A, Kassaye Tessma M, Flink M, Dahlgren A, Schildmeijer K, Ekstedt M. Validation of the patient activation measure in patients at discharge from hospitals and at distance from hospital care in Sweden. BMC Public Health. 2019 Dec 19;19(1):1701. doi: 10.1186/s12889-019-8025-1. PMID 31856796
- [Background] Hibbard JH. Using systematic measurement to target consumer activation strategies. Med Care Res Rev. 2009 Feb;66(1 Suppl):9S-27S. doi: 10.1177/1077558708326969. Epub 2008 Dec 3. PMID 19052169
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Background] Hibbard JH, Greene J, Shi Y, Mittler J, Scanlon D. Taking the long view: how well do patient activation scores predict outcomes four years later? Med Care Res Rev. 2015 Jun;72(3):324-37. doi: 10.1177/1077558715573871. Epub 2015 Feb 24. PMID 25716663
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Hibbard JH, Tusler M. Assessing activation stage and employing a "next steps" approach to supporting patient self-management. J Ambul Care Manage. 2007 Jan-Mar;30(1):2-8. doi: 10.1097/00004479-200701000-00002. PMID 17170632
- [Background] Hosseinzadeh H, Verma I, Gopaldasani V. Patient activation and Type 2 diabetes mellitus self-management: a systematic review and meta-analysis. Aust J Prim Health. 2020 Dec;26(6):431-442. doi: 10.1071/PY19204. PMID 33222755
- [Background] Kinney RL, Lemon SC, Person SD, Pagoto SL, Saczynski JS. The association between patient activation and medication adherence, hospitalization, and emergency room utilization in patients with chronic illnesses: a systematic review. Patient Educ Couns. 2015 May;98(5):545-52. doi: 10.1016/j.pec.2015.02.005. Epub 2015 Feb 19. PMID 25744281
- [Background] Kosar C, Besen DB. Adaptation of a patient activation measure (PAM) into Turkish: reliability and validity test. Afr Health Sci. 2019 Mar;19(1):1811-1820. doi: 10.4314/ahs.v19i1.58. PMID 31149012
- [Background] Lee MK, Lee KH, Yoo SH, Park CY. Impact of initial active engagement in self-monitoring with a telemonitoring device on glycemic control among patients with type 2 diabetes. Sci Rep. 2017 Jun 20;7(1):3866. doi: 10.1038/s41598-017-03842-2. PMID 28634381
- [Background] Lee SWH, Chan CKY, Chua SS, Chaiyakunapruk N. Comparative effectiveness of telemedicine strategies on type 2 diabetes management: A systematic review and network meta-analysis. Sci Rep. 2017 Oct 4;7(1):12680. doi: 10.1038/s41598-017-12987-z. PMID 28978949
- [Background] Lorig K, Ritter PL, Laurent DD, Plant K, Green M, Jernigan VB, Case S. Online diabetes self-management program: a randomized study. Diabetes Care. 2010 Jun;33(6):1275-81. doi: 10.2337/dc09-2153. Epub 2010 Mar 18. PMID 20299481
- [Background] Lorig K, Ritter PL, Villa FJ, Armas J. Community-based peer-led diabetes self-management: a randomized trial. Diabetes Educ. 2009 Jul-Aug;35(4):641-51. doi: 10.1177/0145721709335006. Epub 2009 Apr 30. PMID 19407333
- [Background] McDonnell ME. Telemedicine in Complex Diabetes Management. Curr Diab Rep. 2018 May 24;18(7):42. doi: 10.1007/s11892-018-1015-3. PMID 29797292
- [Background] Melby K, Nygard M, Brobakken MF, Grawe RW, Guzey IC, Reitan SK, Vedul-Kjelsas E, Heggelund J, Lara-Cabrera ML. Test-Retest Reliability of the Patient Activation Measure-13 in Adults with Substance Use Disorders and Schizophrenia Spectrum Disorders. Int J Environ Res Public Health. 2021 Jan 29;18(3):1185. doi: 10.3390/ijerph18031185. PMID 33572717
- [Background] Michaud TL, Siahpush M, King KM, Ramos AK, Robbins RE, Schwab RJ, Clarke MA, Su D. Program completion and glycemic control in a remote patient monitoring program for diabetes management: Does gender matter? Diabetes Res Clin Pract. 2020 Jan;159:107944. doi: 10.1016/j.diabres.2019.107944. Epub 2019 Nov 23. PMID 31765684
- [Background] Michaud TL, Siahpush M, Schwab RJ, Eiland LA, DeVany M, Hansen G, Slachetka TS, Boilesen E, Tak HJ, Wilson FA, Wang H, Pagan JA, Su D. Remote Patient Monitoring and Clinical Outcomes for Postdischarge Patients with Type 2 Diabetes. Popul Health Manag. 2018 Oct;21(5):387-394. doi: 10.1089/pop.2017.0175. Epub 2018 Mar 27. PMID 29583057
- [Background] Moljord IE, Lara-Cabrera ML, Perestelo-Perez L, Rivero-Santana A, Eriksen L, Linaker OM. Psychometric properties of the Patient Activation Measure-13 among out-patients waiting for mental health treatment: A validation study in Norway. Patient Educ Couns. 2015 Nov;98(11):1410-7. doi: 10.1016/j.pec.2015.06.009. Epub 2015 Jun 23. PMID 26146239
- [Background] Norris SL, Lau J, Smith SJ, Schmid CH, Engelgau MM. Self-management education for adults with type 2 diabetes: a meta-analysis of the effect on glycemic control. Diabetes Care. 2002 Jul;25(7):1159-71. doi: 10.2337/diacare.25.7.1159. PMID 12087014
- [Background] Pillay J, Armstrong MJ, Butalia S, Donovan LE, Sigal RJ, Vandermeer B, Chordiya P, Dhakal S, Hartling L, Nuspl M, Featherstone R, Dryden DM. Behavioral Programs for Type 2 Diabetes Mellitus: A Systematic Review and Network Meta-analysis. Ann Intern Med. 2015 Dec 1;163(11):848-60. doi: 10.7326/M15-1400. Epub 2015 Sep 29. PMID 26414227
- [Background] Pressman AR, Kinoshita L, Kirk S, Barbosa GM, Chou C, Minkoff J. A novel telemonitoring device for improving diabetes control: protocol and results from a randomized clinical trial. Telemed J E Health. 2014 Feb;20(2):109-14. doi: 10.1089/tmj.2013.0157. Epub 2014 Jan 3. PMID 24404816
- [Background] Rademakers J, Nijman J, van der Hoek L, Heijmans M, Rijken M. Measuring patient activation in The Netherlands: translation and validation of the American short form Patient Activation Measure (PAM13). BMC Public Health. 2012 Jul 31;12:577. doi: 10.1186/1471-2458-12-577. PMID 22849664
- [Background] Rask KJ, Ziemer DC, Kohler SA, Hawley JN, Arinde FJ, Barnes CS. Patient activation is associated with healthy behaviors and ease in managing diabetes in an indigent population. Diabetes Educ. 2009 Jul-Aug;35(4):622-30. doi: 10.1177/0145721709335004. Epub 2009 Apr 28. PMID 19419972
- [Background] Robson N, Hosseinzadeh H. Impact of Telehealth Care among Adults Living with Type 2 Diabetes in Primary Care: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Int J Environ Res Public Health. 2021 Nov 19;18(22):12171. doi: 10.3390/ijerph182212171. PMID 34831925
- [Background] Sacks RM, Greene J, Hibbard J, Overton V, Parrotta CD. Does patient activation predict the course of type 2 diabetes? A longitudinal study. Patient Educ Couns. 2017 Jul;100(7):1268-1275. doi: 10.1016/j.pec.2017.01.014. Epub 2017 Jan 25. PMID 28159442
- [Background] Salehi S, Olyaeemanesh A, Mobinizadeh M, Nasli-Esfahani E, Riazi H. Assessment of remote patient monitoring (RPM) systems for patients with type 2 diabetes: a systematic review and meta-analysis. J Diabetes Metab Disord. 2020 Jan 10;19(1):115-127. doi: 10.1007/s40200-019-00482-3. eCollection 2020 Jun. PMID 32550161
- [Background] Skolasky RL, Mackenzie EJ, Riley LH 3rd, Wegener ST. Psychometric properties of the Patient Activation Measure among individuals presenting for elective lumbar spine surgery. Qual Life Res. 2009 Dec;18(10):1357-66. doi: 10.1007/s11136-009-9549-0. Epub 2009 Nov 15. PMID 19916057
- [Background] Steinsbekk A, Rygg LO, Lisulo M, Rise MB, Fretheim A. Group based diabetes self-management education compared to routine treatment for people with type 2 diabetes mellitus. A systematic review with meta-analysis. BMC Health Serv Res. 2012 Jul 23;12:213. doi: 10.1186/1472-6963-12-213. PMID 22824531
- [Background] Stellefson M, Dipnarine K, Stopka C. The chronic care model and diabetes management in US primary care settings: a systematic review. Prev Chronic Dis. 2013;10:E26. doi: 10.5888/pcd10.120180. PMID 23428085
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Su D, Michaud TL, Estabrooks P, Schwab RJ, Eiland LA, Hansen G, DeVany M, Zhang D, Li Y, Pagan JA, Siahpush M. Diabetes Management Through Remote Patient Monitoring: The Importance of Patient Activation and Engagement with the Technology. Telemed J E Health. 2019 Oct;25(10):952-959. doi: 10.1089/tmj.2018.0205. Epub 2018 Oct 27. PMID 30372366
- [Background] Sun C, Sun L, Xi S, Zhang H, Wang H, Feng Y, Deng Y, Wang H, Xiao X, Wang G, Gao Y, Wang G. Mobile Phone-Based Telemedicine Practice in Older Chinese Patients with Type 2 Diabetes Mellitus: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jan 4;7(1):e10664. doi: 10.2196/10664. PMID 30609983
- [Background] Tang PC, Overhage JM, Chan AS, Brown NL, Aghighi B, Entwistle MP, Hui SL, Hyde SM, Klieman LH, Mitchell CJ, Perkins AJ, Qureshi LS, Waltimyer TA, Winters LJ, Young CY. Online disease management of diabetes: engaging and motivating patients online with enhanced resources-diabetes (EMPOWER-D), a randomized controlled trial. J Am Med Inform Assoc. 2013 May 1;20(3):526-34. doi: 10.1136/amiajnl-2012-001263. Epub 2012 Nov 20. PMID 23171659
- [Background] Tchero H, Kangambega P, Briatte C, Brunet-Houdard S, Retali GR, Rusch E. Clinical Effectiveness of Telemedicine in Diabetes Mellitus: A Meta-Analysis of 42 Randomized Controlled Trials. Telemed J E Health. 2019 Jul;25(7):569-583. doi: 10.1089/tmj.2018.0128. Epub 2018 Aug 20. PMID 30124394
- [Background] Timpel P, Oswald S, Schwarz PEH, Harst L. Mapping the Evidence on the Effectiveness of Telemedicine Interventions in Diabetes, Dyslipidemia, and Hypertension: An Umbrella Review of Systematic Reviews and Meta-Analyses. J Med Internet Res. 2020 Mar 18;22(3):e16791. doi: 10.2196/16791. PMID 32186516
- [Background] Wubben DP, Vivian EM. Effects of pharmacist outpatient interventions on adults with diabetes mellitus: a systematic review. Pharmacotherapy. 2008 Apr;28(4):421-36. doi: 10.1592/phco.28.4.421. PMID 18363526
- See also: Centers For Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, Division of Population Health. BRFSS Prevalence & Trend Data — https://nccd.cdc.gov/BRFSSPrevalence/rdPage.aspx?rdReport=DPH_BRFSS.ExploreByLocation&rdProcessAction=&SaveFileGenerated=1&irbLocationType=States&islLocation=23&islState=&islCounty=&islClass=CLASS03&islTopic=TOPIC18&islYear=2020&hidLocationType=States&hidLocation=23&hidClass=CLASS03&hidTopic=TOPIC18&hidTopicName=Diabetes&hidYear=2020&irbShowFootnotes=Show&rdICL-iclIndicators=DIABETE4&iclIndicators_rdExpandedCollapsedHistory=&iclIndicators=DIABETE4&hidPreviouslySelectedIndicators=&DashboardColumnCount=2&rdShowElementHistory=divTopicUpdating%3dHide%2cislTopic%3dShow%2cdivYearUpdating%3dHide%2cislYear%3dShow%2c&rdScrollX=0&rdScrollY=99&rdRnd=57890
- See also: Centers for Medicare and Medicaid Services. DM-2 (NQF 0059): Diabetes: Hemoglobin A1c (HbA1c) Poor Control (>9%).; 2019. Accessed January 20, 2022. — https://qpp.cms.gov/docs/QPP_quality_measure_specifications/Web-Interface-Measures/2020_Measure_DM-2_CMSWebInterface.pdf
- See also: International Diabetes Federation. IDF Diabetes Atlas. IDF Diabetes Atlas. Published 2021 — https://diabetesatlas.org/
- See also: Lisa A. States with the biggest rural populations. Stacker. Published April 8, 2019. — https://stacker.com/stories/2779/states-biggest-rural-populations?page=5
- See also: National Clinical Care Commission. Report to Congress on Leveraging Federal Programs to Prevent and Control Diabetes and Its Complications. Department of Health and Human Services; 2021. Accessed January 31, 2022. — https://health.gov/sites/default/files/2022-01/NCCC%20Report%20to%20Congress.pdf